CLINICAL TRIAL: NCT01518725
Title: The Effect of Vitamin D Supplementation on Muscle Power in Elite Cyclist
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oklahoma State University (Other)
Collaborators: Mid America Athletic Training Association (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: ED11189
Record Dates: First submitted 2012-01-18; First posted 2012-01-26 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-04

CONDITIONS: Muscle Power
Keywords: Muscle Power; Vitamin D; Vitamins; Cholecalciferol
MeSH Terms: interventions — Vitamin D; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D Supplementation (Experimental): The vitamin D supplementation will consist of 100 mcg of vitamin D/d, to be taken throughout the day. Participants will achieve 100 mcg by taking 2 x 25 mcg capsules per day. One will be taken at each time point (i.e., morning and evening) throughout the day.
  Interventions: Dietary Supplement: Vitamin D
- Gel-like Substance (Placebo Comparator): Participants in the placebo group will receive a capsule containing the inactive ingredients that include cellulose and silica to create a gel-like substance
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D — The vitamin D supplementation will consist of a capsule of 100 mcg of vitamin D/d, to be taken throughout the day. Participants will achieve 100 mcg by taking 2 x 25 mcg capsules per day. One will be taken at each time point (i.e., morning and evening) throughout the day. They will take the vitamin D supplement for the 6 month intervention period
  Other Names: Cholecalciferol
  Arms: Vitamin D Supplementation
Dietary Supplement: Placebo — Participants in the placebo group will receive a capsule containing the inactive ingredients that include cellulose and silica to create a gel-like substance
  Arms: Gel-like Substance

SUMMARY:
The purpose of this study is to evaluate the change in vitamin D status with the change in muscular strength and muscular power in highly trained athletes over a 9-month study period. The investigators hypothesize that the greatest muscular strength and power gains will be demonstrated in the athletes who achieve and maintain a 25(OH)-D > 50 ng/mL (but < 100 ng/mL) over the 6 month study duration.

This hypothesis will be tested by carrying out the following specific aims: Aim 1. to determine the extent to which increasing serum 25(OH)D to > 50 ng/mL is associated with improved muscular power by assessing specific performance measures (e.g. Vertical Jump Test and Wingate test) relative to lean body mass; and Aim 2. to examine the correlation between vitamin D status and muscular power over time.

DETAILED DESCRIPTION:
Study will be advertised through flyers at the training facilities and by word of mouth. Researchers will schedule meeting with club members at the training facilities. At the meetings, the researchers will give an explanation of the study and address any concerns or questions that they may have. Cyclist will have an opportunity to sign up for participation on a sign-up sheet or e-mail the PI directly to minimize any chance of coercion. Meetings will take place in the training facilities in Tulsa, Oklahoma or the Oklahoma City Metropolitan Area. At this time, subjects will complete an informed consent along with demographic, anthropometric and health history, sunlight exposure, calcium and food frequency questionnaires and PAR Q. All subjects will be asked to fill out the questionnaires in the training facilities at various locations to ensure privacy. After completion of the appropriate questionnaires, cyclist will be have venous blood from the dominant arm (i.e., ~ 5 cc of blood) collected by a licensed medical professional and serum samples stored for future analysis of vitamin D metabolites (i.e., 25-OH-vitamin D and 1,25-OH-vitamin D) and parathyroid hormone (PTH) concentrations. The cyclist's arm will be cleaned with an alcohol swab, the blood will be drawn into a sterile vacutainer using a sterile needle. At the completion of blood collection, the arm will again be cleaned using sterile gauze and covered by a band aid to minimize the risk of infection. Samples will be placed on ice in an ice chest until they are processed in the Nutritional Sciences laboratories at Oklahoma State University. Subjects will then undergo skin tone analyses followed by evaluation of specific performance measures of muscular strength and power. These performance measures include: vertical jump test and a Wingate Power Test. All testing and blood collection will take place at the training facilities.

Within 4 weeks of completing the baseline assessment, the investigators will meet with the cyclist at their training facilities. Participants will be randomly assigned to placebo or the vitamin D supplemented group. The vitamin D supplementation will consist of 100 mcg of vitamin D/d, to be taken throughout the day. Participants will achieve 100 mcg by taking 2 x 25 mcg capsules per day. One will be taken at each time point (i.e., morning and evening) throughout the day. Currently, there is no evidence suggesting that athletes require more vitamin D then the general population for their age. Although we do not anticipate that the dose of vitamin D used in this study, will produce intoxication (150 ng/mL), subjects who exceed 100 ng/ml (i.e., upper end of the normal range) at any time will be asked to discontinue the study. Studies that have demonstrated the benefits of vitamin D supplementation on muscular strength and muscular power have combined vitamin D with calcium. Therefore, all subjects (placebo and vitamin D supplemented group) will be given a commercially available supplement of calcium and instructed to take with breakfast. The calcium supplement is in the form of calcium citrate (500 mg per capsule).

ELIGIBILITY:
Inclusion Criteria:

* Elite Cyclist (level 1,2 or 3)

Exclusion Criteria:

* Currently prescribed vitamin D without physician approval to participate in study
* Participants who respond "yes' to PAR-Q and do not get physician approval to participate in study

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 103 (Actual)
Dates: Start 2012-01; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Change in Vitamin D status from baseline to 3 months and 6 months | Up to 6 months
  Non fasting blood samples will be used for the evaluation of vitamin D metabolites. Venous blood (~5 cc) will be collected from the non-dominant arm by a trained phlebotomist, centrifuged at 2,000 rpm and serum stored at -80° C. Two vitamin D metabolites, 25 (OH) D and 1,25 (OH)2 D and serum PTH will be assessed.
Change in Power Output from baseline to 3 months and 6 months | Up to 6 months
  Power will be assessed using a Vertical Jump Test and a Wingate Power Test.

SECONDARY OUTCOMES:
Sun Exposure Questionnaire | Up to 6 months
  Participants will complete a sun exposure questionnaire (SEQ) to estimate vitamin D synthesis. The SEQ is a 2 point questionnaire that assesses exposure in a week's time period. Sun exposure can be calculated by day and by week. This questionnaire is currently in press.
Skin Tone Measurement | Up to 6 months
  Skin tone will be assessed using the SmartProbe 400 for skin color measurement (IMS, Inc., Portland, ME). The measurement will be performed on the inner and outer portion of the forearm (dominant arm).
Food Frequency Questionnaire | Up to 6 months
  A food frequency questionnaire (FFQ) will estimate dietary vitamin D intake. The FFQ is a 12 point questionnaire that assesses vitamin D supplement usage and the intake of foods that are vitamin D rich.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel A Hildebrand, M.Ed, Principal Investigator — Oklahoma State University; Brenda Smith, PhD, Principal Investigator — Oklahoma State University
Locations (1):
- Oklahoma State University, Stillwater, Oklahoma, United States